CLINICAL TRIAL: NCT02617004
Title: Multicenter Trial Treatment of Philadelphia Chromosome Negative (Ph-) B-lineage Acute Lymphoblastic Leukemia (ALL) of Young Adults (18-59 Years).
Brief Title: Multicenter Trial Treatment of Philadelphia Chromosome Negative B-cell Acute Lymphoblastic Leukemia of Young Adults
Acronym: GRAALL-2014/B
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: AOM12629_3
Record Dates: First submitted 2015-11-25; First posted 2015-11-30 (Estimated); Last update posted 2019-02-19 (Actual); Status verified 2019-02

CONDITIONS: Philadelphia Chromosome Negative Adult B-cell Acute Lymphoblastic Leukemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — leukemic cells, nucleic acids, serum
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to prospectively validate the new risk model, based on minimal residual disease (MRD) response level and oncogenetic status by comparing historical results of GRAALL-2005 with those of GRAALL-2014 in an identical population of patients (Philadelphia chromosome negative, B lineage ALL, aged 18 to 59 years old).

ELIGIBILITY:
Inclusion Criteria:

1. Whose blood and bone marrow explorations have been completed before the steroids prephase
2. Aged 18 to 59 years old with not previously treated (including intrathecal injection) B-lineage-ALL newly diagnosed according to the WHO 2008 definition with ≥ 20% bone marrow blasts
3. Whose karyotype shows no t(9;22) and/or the absence in molecular biology of breakpoint cluster region-Abelson (BCR-ABL)
4. With Eastern Cooperative Oncology Group (ECOG) performance status ≤3
5. With or without central nervous system (CNS) or testis involvement
6. Without other evolving cancer (except basal cell carcinoma of the skin or "in situ" carcinoma of the cervix) or its radiotherapy or chemotherapy treatment should be finished at least since 6 months
7. Having signed a written informed consent
8. With efficient contraception for women of childbearing age (excluding estrogens and IUD)
9. With health insurance coverage
10. Who have received or being receiving the steroid prephase

Exclusion Criteria:

1. With lymphoblastic lymphoma and bone marrow blasts < 20%, Burkitt-type ALL, or with antecedents of chronic myeloid leukemia (CML) or other myeloproliferative neoplasm
2. With contra-indication to anthracyclines or any other general or visceral contra-indication to intensive therapy except if considered related to the ALL:

   * Aspartate transaminase (AST) and/or alanine transaminase (ALT) > 5 x upper limit of normal range (ULN)
   * Total bilirubin ≥ 2.5 x upper limit of normal range (ULN)
   * Creatinine >1.5x upper limit of normal range (ULN) or creatinine clearance <50 mL/mn
3. Myocardial infarction within 6 months prior to inclusion in the trial, cardiomyopathy (NYHA grade III or IV), left ventricle ejection fraction (LVEF) < 50% and or Shortening fraction < 30%,
4. Active severe infection or known seropositivity for HIV or human T cell leukemia/lymphoma virus type 1 (HTLV1) or active hepatitis B or C
5. Pregnant (beta-Human Chorionic Gonadotropin positive) or nursing woman
6. Not able to bear with the procedures or the frequency of visits planned in the trial
7. Unable to consent, under tutelage or curators, or judiciary safeguard.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Young Adults (age 18-59) with Philadelphia Chromosome Negative B-cell Acute Lymphoblastic Leukemia
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2016-02; Primary Completion 2020-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Disease free survival (DFS) | 4 years

SECONDARY OUTCOMES:
Cumulative incidence of relapse (CIR) | 4 years
non relapse mortality (NMR) | 4 years
Overall survival | 4 years
Cumulative incidence of relapse (CIR) after censoring at allo-stem cell transplantation (SCT) in first complete remission (CR) | 4 years
overall survival after censoring at allo-stem cell transplantation (SCT) in first complete remission (CR) | 4 years
Non relapse mortality (NRM) after censoring at allo-stem cell transplantation (SCT) in first complete remission (CR) | 4 years
Disease free survival (DFS) after censoring at allo-stem cell transplantation (SCT) in first complete remission (CR) | 4 years
Minimal residual disease (MRD) | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Hervé Dombret, MDPhD, Principal Investigator — APHP
Locations (1):
- Hématologie Adulte, Saint Louis hospital, Paris, France

REFERENCES:
- [Derived] Boissel N, Chevret S, Rigal-Huguet F, Leguay TT, Hunault M, Graux C, Chalandon Y, Delabesse E, Hicheri Y, Chevallier P, Balsat M, Pastoret C, Escoffre-Barbe M, Pasquier F, Joris M, Thiebaut A, Huynh A, Dhedin N, Lemasle E, Bonmati C, Maury S, Guillerm G, Berceanu A, Schanz U, Cluzeau T, Turlure P, Rousselot P, De Prijck B, Grardel N, Bene MC, Lafage-Pochitaloff M, Cuccuini W, Ifrah NH, Lheritier V, Asnafi V, Clappier E, Dombret H. Age-adapted chemotherapy and MRD-oriented transplant for Ph-negative acute lymphoblastic leukemia: the GRAALL-2014 trial. Blood. 2025 Oct 24:blood.2025029611. doi: 10.1182/blood.2025029611. Online ahead of print. PMID 41135009